CLINICAL TRIAL: NCT03906643
Title: A Phase I Study of HS-201, an HSP90 Inhibitor-linked Verteporfin for Detection of Solid Malignancies
Brief Title: HS-201, an HSP90 Inhibitor-linked Verteporfin for Detection of Solid Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding exhausted
Sponsor: Herbert Lyerly (Other)
Responsible Party: Sponsor-Investigator, Herbert Lyerly, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00102188
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor
Keywords: tumor; verteporfin; HSP90 inhibitor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label phase I study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HS-201 (Experimental): HS-201 will be administered intravenously as a single dose
  Interventions: Drug: HS-201

INTERVENTIONS:
Drug: HS-201 — HS-201 will be administered intravenously as a single dose

SUMMARY:
HS-201 is Verteporfin-tethered HSP90 inhibitor for clinical imaging of selective tumor binding. HS-201 consists of a HSP90 inhibitor that binds competitively to the Hsp90 ATP binding domain connected by a linker to a photosensitizing agent (verteporfin) that can be used for imaging. HS-201 can freely enter tumor cells to selectively bind Hsp90. Due to the the verteporfin, HS-201 accumulation in the malignant cells allows for specific visualization of tumors within the body and verteporfin may allow for photodynamic therapy of tumors.

DETAILED DESCRIPTION:
The product to be tested in this study, HS-201, is a tumor imaging agent.

Hsp90 (heat shock protein 90) is a chaperone protein that aids in the folding, stabilization, and degradation of cellular proteins and is found in virtually all living organisms. Cancer cells in particular have high expression of Hsp90. Hsp90 has three structural domains including an N-terminal domain that contains an ATP binding site. Small molecule inhibitors of HSP90 (Hsp90i) can selectively and competitively to the Hsp90 ATP binding domain. HS-196 consists of a HSP90 inhibitor that binds competitively to the Hsp90 ATP binding domain connected by a linker to a photosensitzing agent (verteporfin) that can be used for imaging. HS-201 can freely enter tumor cells to selectively bind Hsp90. Due to the verteporfine, HS-201 accumulation in the malignant cells allows for specific visualization of tumors within the body.

HS-201 will be used in this investigation for the imaging of solid tumors The objectives of the study are to determine the dose of HS-201 that achieves the greatest ratio of tumor to normal tissue fluorescence in patients with malignancy, the safety of HS-201 administration in patients with malignancy, the average radiant efficiency in resected tumors following HS-201 administration, the localization of the HS-201 by microscopy of tumor slices, and the PK metrics of HS-201 when administered to patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solid malignancy, stage I-IV.
* Planned surgical resection or biopsy of a malignancy
* ECOG 0 or 1
* Estimated life expectancy > 3 months
* Age ≥ 18 years
* Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5, PTT <1.5X ULN
* Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal or if liver metastases are present < 5 x upper limit of normal.
* Female patients must be of non-child-bearing potential or use effective contraception
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board's guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up, as required by this protocol.

Exclusion Criteria:

* Serious chronic or acute illness considered by the P.I. to constitute an unwarranted high risk for investigational drug treatment.
* Patients with porphyria or a known hypersensitivity to any component of this preparation are excluded.
* Medical or psychological impediment to probable compliance with the protocol.
* Asthma under medical management
* Uncontrolled high blood pressure
* Presence of a known active acute or chronic infection including HIV or viral hepatitis (Hepatitis B and C)).
* Pregnant or nursing women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Fluorescence | 1 day
  Ratio of tumor to normal tissue fluorescence

SECONDARY OUTCOMES:
Number of AEs | 1 month
  Safety of HS-201 administration in patients with malignancy
Radiant Efficiency | 1 day
  The average radiant efficiency in resected tumors following HS-201 administration
HS-201 Localization | 1 week
  Localization of the HS-196 by microscopy of tumor slices
Maximum Plasma concentration Cmax | 1 week
  PK metrics of HS-201 when administered IV to patients

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No